CLINICAL TRIAL: NCT00707928
Title: Intravenous Nitroglycerin for Retained Placenta Extraction: a Multicenter Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Shusee Visalyaputra, Mahidol University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si249/2007
Record Dates: First submitted 2008-06-28; First posted 2008-07-01 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2008-06

CONDITIONS: Retained Placenta
Keywords: retained placenta
MeSH Terms: conditions — Placenta, Retained | interventions — Nitroglycerin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 1=nitroglycerine 100 microgram intravenous100-200 microgram of IV.
  Interventions: Drug: nitroglycerine
- 2 (Placebo Comparator): 2=placebo with the same volume as NTG 100-200 microgram of IV.
  Interventions: Other: NSS

INTERVENTIONS:
Drug: nitroglycerine — nitroglycerine 100 microgram intravenous.Once the placenta had been delivered, oxytocin or ergometrine will be administered. Fentanyl 50-100 microgram can be given if the cord traction is considered painful.
  Other Names: trinitroglycerin,trinitroglycerine,glyceryl trinitrate
  Arms: 1
Other: NSS — NSS.Once the placenta had been delivered, oxytocin or ergometrine will be administered. Fentanyl 50-100 microgram can be given if the cord traction is considered painful.
  Other Names: normal saline
  Arms: 2

SUMMARY:
Primary objective The primary objective of this study is to see whether intravenous (IV) NTG 100-200 microgram can effectively help extract retained placenta as compared to placebo, in a randomized controlled multicenter study.

Secondary objective is to compare the hypotensive effects of NTG as compared to placebo, including others side effects such as headache, blood loss, or others.

DETAILED DESCRIPTION:
After the approval of the Ethical committee of each institute, and consent signed by the patient, 100 patients with retained placenta were divided into 2 groups in 5 tertiary care centers, university hospitals. By using the program research randomizer (from www. Randomizer.org/form.htm), with the block of 10 and the numbers within the concealed envelopes, totally 100 patients with retained placenta will be divided into 2 groups to have either 100-200 microgram of IV, NTG or IV placebo. Due to unequal number of the cases enrolled in each centers, they will receive 10 envelopes for 10 cases (5 NTG and 5 placebo) at a time. When they finish the first 10 cases, they will start another 10 cases of the next set until all 10 sets has been started. Each of 5 centers might enroll the cases between 10 to 40 cases up to their populations..

Once a diagnosis of retained placenta has been made ( ≥ 30 min after delivery), Hematocrit will be checked and IV crystalloid solution 500 ml has been rapidly perfuse and noninvasive monitored included pulse oximetry, electrocardiogram and noninvasive blood pressure will be monitored.

Patients with signs of hypovolemia ( SBP < 100 mmHg, or pulse > 100/min), or ASA classification > II will be excluded from the study.

First step: In the treatment group, 100 microgram of NTG will be given and wait for 80 seconds ( maximum relaxation effects of IV NTG)(5,6) before starting gently cord traction (1min). If the placenta can not be extracted, another 100 microgram NTG from the same syringe will be given and wait for another 80 seconds before starting another extraction (1min), If the placenta can not be extracted, it will be considered failed. In the placebo group, NSS will be used instead of NTG.

Second step: To give a chance for patients in placebo group, another syringe with 200 microgram will be given as in the first step for the placebo group. In the treatment group, NSS will be used instead of NTG. The outcome in the second step will not be included in the first step.( The solutions in both syringes which will be prepared by the research assistant who will not involve in the study, will be blinded to the patient, the obstetrician, the anesthesiologist and the investigator) General anesthesia will be used for manual removal of placenta in cases that placenta can not be extracted after the second step.

Once the placenta had been delivered, oxytocin or ergometrine will be administered. Fentanyl 50-100 microgram can be given if the cord traction is considered painful.

Vital signs will be recorded before the first NTG bolus and thereafter at 1 min interval for 5 min then every 2 min for 10 min then every 5 min. for 20 min(see the CRF).

The patient will be followed up closely for 24 h postoperatively and Hct will be checked , including the final results upon discharge home.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant patient (ASA classification I ,II )
* Normal pregnancy with at least 28 week gestation

Exclusion Criteria:

* ASA classification III and up
* Having complication of pregnancy such as hypertensive disease of pregnancy,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
successful of placenta extraction | 5 mintues

SECONDARY OUTCOMES:
hypotension | 20 mintues
headache | 2 hour
blood loss | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Shusee Visalyaputra, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok 10700
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Bangkok, Thailand